CLINICAL TRIAL: NCT00220441
Title: Cognitive Effects of Aerobic Exercise for Adults With Impaired Glucose Tolerance: A Controlled Trial
Brief Title: Cognitive Effects of Aerobic Exercise for IGT Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: American Diabetes Association (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDIS 0009; ADA BL19 (SIBCR)
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Impaired Glucose Tolerance
Keywords: IGT; exercise; cognition; insulin; aging; aerobic
MeSH Terms: conditions — Glucose Intolerance; Motor Activity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Aerobic exercise

SUMMARY:
The specific aims for the study will be to determine if aerobic exercise enhances cognition for older adults who are at risk for developing type II diabetes mellitus (T2DM), and to evaluate whether change in insulin sensitivity predicts cognitive performance for subjects randomized to the aerobic exercise group. Sedentary older adults diagnosed with impaired glucose tolerance using an oral glucose tolerance test will participate in a 6-month supervised protocol of either aerobic exercise or stretching. Cognitive testing and blood collection will occur at baseline, and months 3 and 6. Before and after the 6-month intervention, insulin sensitivity, maximum aerobic capacity, and body fat composition and distribution (via CT scan) will be assessed for all subjects. The results of this study may provide support for a relatively simple and inexpensive treatment strategy that specifically targets many of the health factors that directly influence risk of cognitive decline associated with T2DM for older adults.

DETAILED DESCRIPTION:
The benefits of exercise on cognition have been demonstrated both in animals and humans. Exercise has salutary effects on glucoregulation and visceral adiposity, an important link for adults with impaired glucose tolerance (IGT) and type 2 diabetes mellitus (T2DM). Exercise also upregulates neurotrophic activity, an effect that serves to increase neuronal viability in the same brain regions that support complex cognitive functions affected by metabolic disease. In this proposed controlled intervention trial, the hypothesis is that aerobic exercise will have a beneficial effect on cognition and several biomarkers that index disease progression for older adults with IGT. 40 older subjects (age: >55 yrs) with IGT, confirmed by OGTT, will be randomized to an aerobic fitness or stretching program for 6 months. Cognitive measures and fasting blood samples will be obtained at baseline, month 3, and month 6. Cognitive tests will evaluate abilities affected by age and by significant glucoregulatory dysregulation. In addition, all subjects will undergo a hyperinsulinemic-euglycemic clamp protocol, a cardiopulmonary fitness assessment, and body fat quantification procedures, immediately before and after the intervention. The specific aims of the study will be to determine if aerobic exercise enhances cognition for older adults with IGT, to evaluate whether exercise-induced change in insulin sensitivity predicts cognitive performance, and to relate exercise effects on insulin sensitivity and cognition to changes in specified biomarkers. The results of this study may provide support for a relatively simple and inexpensive treatment strategy that targets many of the health factors that influence risk of cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with IGT using OGTT, at least 55 years old, sedentary (elevated HR & SOB < 3x/wk for <30min each occasion), good overall health, willing to exercise at least 4 days/week for 6 mos

Exclusion Criteria:

* Significant neurologic disease that might affect cognition, such as AD, stroke, Parkinson's disease, multiple sclerosis, or severe head injury with loss of consciousness; significant medical illness or organ failure, such as liver disease, significant elevations in liver function tests, kidney disease, and uncontrolled hypertension (BP > 140/90 on medication); cardiovascular disease defined as any acute cardiovascular abnormality, such as new or unstable angina, uncontrolled irregular heart beat (treated a-fib and occasional PVC's are OK) or symptomatic heart failure, acute shortness of breath for any reason, or clinically significant edema; chronic lung disease, (COPD/emphysema); musculoskeletal impairment (impaired walking); current use of anti-psychotic, anti-convulsant, anti-coagulant, sedative medication, or cognition-enhancing medications; current or previous use of hypoglycemic agents or insulin.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-07; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change in cognitive scores
Change in insulin sensitivity

SECONDARY OUTCOMES:
Change in biomarkers assayed from blood
Correlation between cognitive scores, insulin sensitivity, biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Laura D. Baker, PhD, Principal Investigator — VA Puget Sound Health Care System; University of Washington
Locations (2):
- United States (2):
  - Veterans Affairs Puget Sound Health Care System, Seattle, Washington
  - Veterans Affairs Puget Sound Health Care System, Tacoma, Washington

REFERENCES:
- [Derived] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Cholerton BA, Plymate SR, Fishel MA, Watson GS, Duncan GE, Mehta PD, Craft S. Aerobic exercise improves cognition for older adults with glucose intolerance, a risk factor for Alzheimer's disease. J Alzheimers Dis. 2010;22(2):569-79. doi: 10.3233/JAD-2010-100768. PMID 20847403